CLINICAL TRIAL: NCT04296448
Title: Evaluation of Cellphone Based Otoscopy in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00187508
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Ear Infection; Pediatric Disease; Acute Otitis Media
Keywords: cellscope; mobile device; pediatric trainees; acute otitis media; ear infection
MeSH Terms: conditions — Otitis; Otitis Media

STUDY DESIGN:
Intervention Model Description: Block randomization, pediatric trainees are exposed in 2-week blocks: 1 week with Cellscope available, 1 week with the traditional otoscope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Otoscope (No Intervention): Pediatric trainees use a traditional otoscope to evaluate pediatric patient ears. Trainees' supervisors will also evaluate patients with the traditional otoscope. The study evaluates concordance of the exams.
- Cellscope (Experimental): Pediatric trainees use a cellphone otoscope (Cellscope) to evaluate pediatric patient ears. Trainees' supervisors will evaluate patients remotely with the video on the cellphone otoscope. The study evaluates concordance of the exams.
  Interventions: Device: Cellscope

INTERVENTIONS:
Device: Cellscope — Cellphone otoscope (Cellscope) to evaluate pediatric patient ears.
  Arms: Cellscope

SUMMARY:
The Cellscope is an iPhone-based otoscope that uses the iPhone camera and light source to capture HIPAA compliant images and video recordings of the external and middle ear structure. This technology allows multiple providers, at different levels of training, the ability to simultaneously exam a child's external and middle ear structures. The investigators hypothesize this device will result in improved concordance in trainee/supervisor exam findings, increase trainee confidence in exam findings, decreased antibiotic prescriptions, and fewer repeat exams by multiple providers. Thus, this study has the potential to improve physician training and examination confidence, decrease the unnecessary use of antibiotics, and improve the patient/caregiver experience in healthcare interactions.

DETAILED DESCRIPTION:
Abstract

Concerns about middle and external ear infections and discomfort are frequent chief complaints that bring children to pediatric providers. On top of this, there are numerous non-ear complaints (e.g. head trauma) that warrant a complete evaluation of the middle and external ear structures. At present, the middle and external ear is examined with standard direct otoscopy, commonly using a handheld otoscope. Otoscopy is defined as the visualization of the external and middle ear structures, including the tympanic membrane, ossicles, middle ear fluid, ear canal, etc. The skill of otoscopy is taught early in the medical trainees' career, most often in the first or second year of medical school. This skill is further honed during the pediatric medical student clerkship and pediatric residency, however there is not an efficient and patient-centered mechanism for direct visualization and teaching of trainees. Because of this, it is nearly impossible for trainees to receive feedback on trainees' visualization and interpretation skills. Based on the investigators' experience, trainee exams are often not repeated by clinical supervisors as the trainees progress in training. When supervisors do repeat ear exams (i.e., trainee is uncertain of findings), it is challenging to determine if the trainee fully appreciates exam findings. Ear exam findings directly inform the clinical decision-making (e.g., prescribing antibiotics for acute otitis media (AOM)) and uncertainty often results in unnecessary prescribing.

Objectives

Aim 1: To establish whether a smartphone otoscope improves diagnostic accuracy of tympanic membrane (TM) pathology for trainees, compared to supervisor.

Aim 2: To determine whether smartphone otoscope improves diagnostic confidence of trainees, thereby reducing frequency of antibiotic prescriptions for AOM.

Aim 3: To determine whether there is a change in repeat exam rates by supervisors, comparing with/without Cellscope.

Aim 4: To determine whether trainees convert to traditional otoscope use during the weeks that Cellscope is available.

ELIGIBILITY:
Inclusion Criteria:

* All trainees and supervisors
* All patients where otoscopy would traditionally be indicated, at the discretion of the clinical team

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Therese Canares, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Children's Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Traditional Otoscope | Cellscope
Started | 98 | 99
Completed | 98 | 99
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Traditional Otoscope | Cellscope | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Customized [Count of Participants; unit: Participants]
  21 years and younger | 98 | 99 | 197
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not collected from any participant.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 99 | 197

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Trainee and Supervisor Utilizing the OMgrade Scale as Assessed by the Concordance-statistic
Description: Concordance of trainee and supervisor utilizing the OMgrade scale, between traditional otoscope and cellscope. Concordance is determined by the concordance-statistic (0-1) in a logistic regression model. The closer the number is to 1 the higher the concordance.
Time Frame: 6 months
Population: 2 subjects were excluded from analysis due to incomplete surveys in the traditional otoscope arm, and 7 from the cell scope arm.
Measure: Number (95% Confidence Interval); unit: concordance-statistic
Arm/Group | Traditional Otoscope | Cellscope
Number analyzed (Participants) | 96 | 92
concordance-statistic | 0.64 [0.57 to 0.70] | 0.75 [0.69 to 0.81]

2. Secondary Outcome: Interrater Reliability as Assessed by a Kappa Statistic
Description: Kappa statistic (Fleiss' Kappa) of trainee and supervisor utilizing the OMgrade scale. The kappa statistic ranges from 0-1. The closer the number is to 1 the higher the agreement.
Time Frame: 6 months
Population: 2 subjects were excluded from analysis due to incomplete surveys in the traditional otoscope arm, and 8 from the cell scope arm.
Measure: Number (95% Confidence Interval); unit: Fleiss' Kappa
Arm/Group | Traditional Otoscope | Cellscope
Number analyzed (Participants) | 96 | 91
Fleiss' Kappa | 0.37 [0.24 to 0.51] | 0.67 [0.57 to 0.78]

3. Secondary Outcome: Number of Patients Who Receive Antibiotics
Description: Number of patients who receive antibiotics between traditional otoscope and cellscope.
Time Frame: 6 months
Population: 2 subjects were excluded from analysis due to incomplete surveys in the traditional otoscope arm, and 6 from the cell scope arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Otoscope | Cellscope
Number analyzed (Participants) | 96 | 93
Participants | 21 | 11

4. Secondary Outcome: Number of Participants Who Receive a Repeat Examination
Description: Number of participants who receive a repeat examination between traditional otoscope and cellscope.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Traditional Otoscope | Cellscope
Number analyzed (Participants) | 96 | 92
Participants | 94 | 25

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Traditional Otoscope | Cellscope
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/99
Other Adverse Events (participants affected / at risk) | 0/98 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT04296448/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/48/NCT04296448/ICF_001.pdf